CLINICAL TRIAL: NCT06854653
Title: An Open-Label, Phase 2 Study of PTX-100 Monotherapy in Patients With Relapsed or Refractory Cutaneous T-Cell Lymphoma.
Brief Title: A Phase 2 Study of PTX 100 in Patients With Relapsed/Refractory CTCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prescient Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTX-100-02-2024
Record Dates: First submitted 2025-02-18; First posted 2025-03-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: CTCL
Keywords: Relapsed or refractory Cutaneous T Cell Lymphoma; CTCL; PTX-100; Mycosis Fungoides; Sezary Syndrome; T Cell Lymphoma; Non-Hodgkin Lymphoma; Cutaneous Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: Randomised parallel recruitment into 2 treatment arms, 500mg/m2 and 1000-mg/m2 for Phase 2a.
  Phase 2b will be non-randomised and are single arm treatment group. The recommended optimal dose which was determined in Phase 2a will be used in Phase 2b.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 2a PTX-100 500mg/m2 (Experimental): Phase 2a PTX-100 will be 500mg/m2 IV infusion over 60 minutes on days 1 to 5 of a 14-day cycle for 4 cycles. This is then followed by IV infusion over 60 minutes on days 1 to 5 of a 21-day cycle for up to 18months.
  Interventions: Drug: PTX-100
- Phase 2a PTX-100 1000mg/m2 (Experimental): Phase 2a PTX-100 will be 1000mg/m2 IV infusion over 60 minutes on days 1 to 5 of a 14-day cycle for 4 cycles. This is then followed by IV infusion over 60 minutes on days 1 to 5 of a 21-day cycle for up to 18months.
  Interventions: Drug: PTX-100
- Phase 2b PTX-100 Recommended Optimal Dose (ROD). (Experimental): Phase 2b PTX-100 will be the Recommended Optimal Dose form Phase 2a and follow the same infusion timeline outlined previously. IV infusion of RD over 60 minutes on days 1 to 5 of a 14-day cycle for 4 cycles then followed by IV infusion of RD over 60 minutes on days 1 to 5 of a 21-day cycle up to 18months.
  Interventions: Drug: PTX-100

INTERVENTIONS:
Drug: PTX-100 — Peptidomimetic inhibitor of GGTase 1

SUMMARY:
This is an open-label, phase 2 randomized study to evaluate the efficacy, safety, pharmacokinetics (PK) and pharmadynamics (PD), of PTX-100 monotherapy at 500 or 1000 mg/m2 in patients with relapsed/refractory Cutaneous T-Cell Lymphoma (CTCL).

PTX-100 will be administered by IV infusion over 60 minutes on days 1 to 5 of a 14-day cycle for 4 cycles, then 21 day cycle thereafter. Subjects will be treated or followed up, if subjects discontinue treatment, for up to 18 months.

DETAILED DESCRIPTION:
PTX-100 from a Phase I study shown to help some CTCL patients. This Phase II study will be conducted in a larger population size and there will be initially two groups/arms in the first phase called Phase 2a. This phase will randomize and enroll 20 subjects into the 500 mg/m2 and 20 subjects into the 1000 mg/m2 PTX treatment arms. After determining the recommended optimal dose from phase 2a, for Phase 2b, 75 subjects will then be allocated into this single arm part of the study.

Once subject has signed the informed consent, subject will undergo a 28 day screening period, where eligibility would be determined. Once subject is eligible, subject will be dosed with IP. Safety bloods will be taken on the first day of every cycle. Pharmacokinetics (PKs) which are blood samples sent to the Sponsors associated laboratory and will be analysed on how PTX-100 interacts biologically. PKs will be taken on Cycle1Day1(C1D1) to C1D5 and C1D8 for the first 4 cycles. Subject will also undergo skin evaluation and safety exams at every Cycle Day 1. Subjects will also complete quality of life questionnaires at every Cycle Day1. Subjects will be on the study for 18months, until disease progression, unacceptable toxicity, participant or Investigator decision, or until study treatment discontinuation criteria are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ≥18 years of age at the time of signing the informed consent.
2. Patient is capable of giving adequate signed informed consent
3. Have a confirmed diagnosis of CTCL with histological confirmation
4. Patients must have greater than or equal to Stage Ib disease.
5. Has received and failed (or intolerant of) at least 2 prior lines of prior systemic therapy for their disease.
6. Has measurable disease defined by at least one of the following, within 28 days prior to start of study treatment: by evaluable by mSWAT or quantifiable by flow cytometry or morphology in blood or measurable by Lugano Criteria.
7. On a stable dose of systemic corticosteroid (< 10 mg prednisone or equivalent) are permitted. Participants on a stable dose of topical corticosteroids are permitted.
8. Washout period- must be 2 weeks (4 weeks for monoclonal antibodies) or 5 -half-lives (whichever is longer) since any prior anti-cancer therapy.
9. Must be human T-cell lymphotropic virus type 1 (HTLV1) negative.
10. Has an ECOG PS of 0 to 2.
11. Life expectancy of 3 months or greater
12. Has adequate bone marrow function.
13. Has adequate hepatic function.
14. Has adequate Renal function.
15. Has adequate coagulation function.
16. Patients with Human Immunodeficiency virus (HIV) must be on established and stable effective anti-retroviral therapy for at least 4 weeks and have an HIV viral load of less than 400 copies/mL.
17. Male patients are eligible to participate if they agree to use a highly effective contraception during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period.
18. Female patients are eligible to participate if they are not pregnant, not breastfeeding, and at least one of the following conditions applies:

    -Not a woman of childbearing potential (WOCBP).
    * OR
    * A WOCBP who agrees to use a contraceptive method that is highly effective (with a failure rate of < 1% per year) or be abstinent from heterosexual intercourse as their preferred method and usual lifestyle, beginning the time of informed consent, during the treatment period and for at least 3 months after the last dose of study treatment.
19. A WOCBP must have a negative serum pregnancy within 72 hours of the first dose of study treatment.
20. Must be willing and able to adhere to the study as judged by the Investigator.

Exclusion Criteria:

1. Patients with known central nervous system involvement.
2. Patients who require the use of strong inhibitors or inducers of CYP enzymes or transporters (e.g., CYP3A4, 2D6, 2C19) or (P-gp, BCRP, OATP1B1, OATP1B3, OAT1. OAT3, OCT2, MATE1 and MATE2-K). Patients who are receiving these medications at Screening can be enrolled into the trial if they discontinue them for at least 14 days or 5 half-lives, whichever is longer, before they commence PTX-100. An alternative pharmacological treatment should be instituted by the treating clinician based on clinical judgement.
3. Significant cardiovascular disease. A history of, or concurrent interstitial lung disease or severely impaired lung function.

5. Active viral, bacterial, fungal infection or other serious infection requiring ongoing systemic treatment. Routine antimicrobial prophylaxis is permitted.

6. Medical history of another malignant tumor within the past 5 years. Exceptions are patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ who have undergone curative therapy with no evidence of disease.

7. On an immunomodulatory drug for concomitant or intercurrent conditions or who have received any of these agents within 4 weeks of baseline.

8. Patients with active viral (any etiology) hepatitis are excluded. However, patients with serologic evidence of chronic hepatitis B virus (HBV) infection (defined by a positive hepatitis B surface antigen test and a positive anti-hepatitis core antigen antibody test) who have a viral load below the limit quantification (HBV deoxyribose nucleic acid titer < 1000 cps/mL or 200 IU/mL) and are not currently on viral suppressive therapy may be eligible and should be discussed with the Medical Monitor. Patients with a history of hepatitis C virus infection who have completed curative antiviral treatment and have a viral load below the limit of quantification may be eligible and should be discussed with the Medical Monitor.

9. A history or current evidence of any condition, laboratory abnormality or other circumstance that might confound the results of the study or interfere with patient participation for the full duration of the study.

10. Prior allogeneic or autologous hematopoietic transplantation 11. Has a known psychiatric disorder that would interfere with compliance with the requirements of the study.

12. Is a consumer of illicit or recreational drugs or has a recent history (within the last year) of drug or alcohol abuse or dependence that in the judgment of the Investigator, would interfere with compliance with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of PTX-100 as determined by ORR. | 18 months from day of first treatment until disease progression, unacceptable toxicity, participant or Investigator decision.
  Objective response rate (ORR): ORR is defined as the proportion of patients who achieved CR or PR as their best response

SECONDARY OUTCOMES:
To further characterize the efficacy of PTX-100 | Within 18 months after PTX-100 initial dose.
  Skin response as per Modified Severity-Weighted Assessment Tool (mSWAT). The mSWAT uses body surface area in 12 body areas to calculate involvement. A weighting factor is also used: Patches, which are flat, earned a multiplier of one. Plaques, which are raised, earned a multiplier of two. Tumors, which are larger and solid, earned a multiplier of three. Lesion BSA multiplied with the weighting factor with the sum of regions affected gives a final mSWAT score.
  The SWAT result is a number is monitored over time. A stable number suggested a stable condition. A lower number suggested less active CTCL and conversely, a higher number suggested more active CTCL.
Progression-free survival (PFS) | Within 18 months after PTX-100 initial dose.
  Defined as the time from the date of PTX-100 initiation to the date of first documented progression or death.
Time to response (TTR) | Within 18 months after PTX-100 initial dose.
  TTR: defined as the time from the date of PTX-100 initiation to first confirmed objective response (CR or PR)
Overall survival (OS) | Within 18 months after PTX-100 initial dose.
  OS: defined as the time interval between the date of PTX-100 initiation and the date of death due to any cause
Duration of response (DoR) | Within 18 months after PTX-100 initial dose.
  DoR: defined as the time interval between the first confirmed objective response (CR or PR) and the first occurrence of objective progression (PD) or death from any cause.
Complete response rate (CRR) | Within 18 months after PTX-100 initial dose.
  Complete response rate (CRR) evaluated according to the Lugano2014 criteria.
Pharmacokinetics (PK) of PTX-100: Cmax | Cycle 1: Day 1 and Day 5: pre-dose, 5 mins post-infusion, and at 1, 2, 4, 6, and 8 hours after dose. Day 2, 3 and 4: 24 hours after previous dose, bloods taken at Pre and at 5 mins post-infusion. Day 8; 72 hours after the Day 5 dose and prior to dosing.
  PTX-100 peak plasma concentration (Cmax) in plasma
Pharmacokinetics (PK) of PTX-100: Tmax | Cycle 1: Day 1 and Day 5: pre-dose, 5 mins post-infusion, and at 1, 2, 4, 6, and 8 hours after dose. Day 2, 3 and 4: 24 hours after previous dose, bloods taken at Pre and at 5 mins post-infusion. Day 8; 72 hours after the Day 5 dose and prior to dosing.
  Time to peak drug concentration in plasma (Tmax)
Pharmacokinetics (PK) of PTX-100: Cmin | Cycle 1: Day 1 and Day 5: pre-dose, 5 mins post-infusion, and at 1, 2, 4, 6, and 8 hours after dose. Day 2, 3 and 4: 24 hours after previous dose, bloods taken at Pre and at 5 mins post-infusion. Day 8; 72 hours after the Day 5 dose and prior to dosing.
  Cmin for the minimum blood plasma concentration reached by PTX-100 during the time interval between administration of two doses
Pharmacokinetics (PK) of PTX-100: AUCtau | Cycle 1: Day 1 and Day 5: pre-dose, 5 mins post-infusion, and at 1, 2, 4, 6, and 8 hours after dose. Day 2, 3 and 4: 24 hours after previous dose, bloods taken at Pre and at 5 mins post-infusion. Day 8; 72 hours after the Day 5 dose and prior to dosing.
  AUCtau, area under the curve from time 0 to time tau (the dosing interval) at steady state. AUCtau is typically expressed in units of concentration multiplied by time (e.g., ng·h/mL)

OTHER OUTCOMES:
To evaluate the effects of Health-related Quality of Life (QoL) | From Baseline till end of study
  To collect the health related questionnaire for CTCL whihc includes Functional Assessment of Cancer Therapy -General (FACT-G), Skindex-29, European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) and ItchyQoL
Exploratory Biomarkers | From Baseline till end of study
  Assessing Biomarker downstream signature of PTX-100 treatment: measurement value (and the change from baseline and throughout the study) of gene/ protein expression in blood samples for each subject using Olink Explore HT high-throughput platform

CONTACTS AND LOCATIONS:
Locations (15):
- United States (6):
  - City of Hope Comprehensive Cancer Cente, Duarte, California
  - University of California Irvine, Irvine, California
  - Yale Cancer Center, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Rochester Skin Lymphoma Medical Group. PLLC, Rochester, New York
  - Virginia Commonwealth University Massey Comprehensive Cancer Cente, Richmond, Virginia
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Epworth Healthcare, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- France (3):
  - CHU de Bordeaux - Hopital Saint André, Bordeaux, Bordeaux
  - Hopital Lyon Sud, Lyon, Pierre-Benite
  - Hopital Saint Louis, Paris, Île-de-France Region
- Italy (3):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna - Policlinico S. Orsola-Malpighi, Bologna, Bologna
  - Universita degli Studi Di Brescia-Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia, Brescia
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan, Milano

IPD SHARING:
Plan to Share IPD: No